CLINICAL TRIAL: NCT02724514
Title: Multi-Parametric Assessment of Breast Lymphedema
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: UHN REB 14-8503-C
Record Dates: First submitted 2015-03-02; First posted 2016-03-31 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer; Breast Lymphedema
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: non-invasive image & bioimpedance based techniques — Ultrasound scans, bioimpedance measurements, clinical photographs and questionnaires will be performed before and after the massage.

SUMMARY:
Breast lymphedema (swelling due to fluid) is a common complication of breast cancer therapy. Unlike lymphedema in the arm, breast lymphedema is not as well-known and has not been studied. At present, no objective and standardized tools exist to evaluate breast lymphedema.

The purpose of this study is to investigate the use of ultrasound analysis and bio-impedance to determine if it is possible to measure the extent of the fluid in the breast.

DETAILED DESCRIPTION:
Breast lymphedema (swelling due to fluid) is a common complication of breast cancer therapy. Limited research has been conducted on the frequency of breast lymphedema with most studies reporting the incidence as ranging from 33 to 48%. Women with breast lymphedema describe breast fullness, heaviness and pain associated with breast swelling and changes that impacts how the breast looks (cosmesis) and also impacts their quality of life.

At present, no objective and standardized tools exist to evaluate breast lymphedema and correlate it with tissue fluid and fibrosis, and their relationships to local symptoms, cosmesis and quality of life.

The goal of the study is to assess and compare photographic, ultrasound and the breast composition in newly diagnosed breast lymphedema, and to assess the use of breast massage to manage breast lymphedema. Developing non-invasive image-based methods may enable researchers to map the extent of lymphedema, monitor its progression and evaluate therapies. This may allow for improved quantitate measures to be undertaken to better assess future strategies intended to prevent or improve the management of this treatment complication.

Patients participating in this study will have ultrasound scans before and after the massage. They will also be asked to complete a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 y/o
* Diagnosis of lymphedema involving the breast
* Diagnosis of in-situ or invasive breast cancer
* Female patients following breast conserving therapy and radiotherapy
* Spoken and written fluency in English; and
* Able to provide informed consent

Exclusion Criteria:

* Pacemaker or implanted stimulator or other contraindication to bioimpedance analysis
* Prior breast surgery on the contra lateral breast
* Presence of active cellulitis within the breast, trunk or arm and
* Presence of active cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast lymphedema Cancer patients with lymphedema
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
Measure Mid-Band Fit (MBF) in normal tissue controls and the corresponding regions of lymphedema | 2 years
  The MBF, measured in dB, is a quantitative ultra-sound (QUS) image parameter used to characterize tissue microstructure
Measure Acoustic Scatterer Diameter (ASD) in normal tissue controls and the corresponding regions of lymphedema | 2 years
  The ASD, measured in mm, is a quantitative ultra-sound (QUS) image parameter used to characterize tissue microstructure

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dinniwall, MD, Principal Investigator — UHN
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada